CLINICAL TRIAL: NCT04268082
Title: The Effects of Insole-based Visual Biofeedback on Weight-bearing in Patients Undergoing Total Hip Replacement. A Randomised Controlled Trial.
Brief Title: Insole-based Visual Biofeedback for Weight-bearing in Total Hip Replacement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pavia (Other)
Responsible Party: Principal Investigator, Luca Marin, Principal Investigator, University of Pavia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20180036031
Record Dates: First submitted 2020-02-06; First posted 2020-02-13 (Actual); Last update posted 2020-02-13 (Actual); Status verified 2020-02

CONDITIONS: Total Hip Replacement; Visual Biofeedback; Weight Bearing

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): The Experimental Group followed the training wearing sensorized insoles that provided plantar pressures and shift of foot center of pressure images reported on monitors.
  Interventions: Device: Visual biofeedback with the use of sensorized insoles
- Control Group (Active Comparator): The Control Group followed verbal instructions of physiotherapist during training.
  Interventions: Other: Standard rehabilitation based on physiotherapist's verbal instructions

INTERVENTIONS:
Device: Visual biofeedback with the use of sensorized insoles — Between the 4th and the 10th day post surgery, both groups performed the same rehabilitation protocol. The experimental group was re-educated to the correct gait dynamics by wearing the sensorized insoles and by using a specific software's graphical interface as a visual biofeedback.
  Arms: Experimental Group
Other: Standard rehabilitation based on physiotherapist's verbal instructions — Between the 4th and the 10th day post surgery, both groups performed the same rehabilitation protocol.The Control group did not wear the insoles, but it carried out the rehabilitation programme under the physiotherapist supervision and with his verbal feedbacks.
  Arms: Control Group

SUMMARY:
The study investigates the effects of visual biofeedback, based on a sensorized system for the dynamic evaluation of the plantar pressure versus rehabilitation with traditional verbal instructions of the physiotherapist, on weight bearing distribution in patients who underwent first total hip replacement. The study is a randomized controlled trial, with parallel groups, without blinding.

DETAILED DESCRIPTION:
Forty patients, who underwent first total hip replacement surgery were enrolled and divided into two groups on second postoperative day. Experimental group followed the training wearing sensorized insoles that provided plantar pressures and shift of foot center of pressure images on three monitors. Control Group followed verbal instructions of physiotherapist during training. From 4th to 10th postoperative day both groups followed the same rehabilitation program including exercises to restore correct weight bearing.

ELIGIBILITY:
Inclusion Criteria:

* 75 ≤ years of age,
* absence of conditions that could alter the gait cycle,
* absence of conditions that could reduce or alter visual ability,
* etherometry ≤ 0.5 mm
* Mini-Mental State Examination (MMSE) score ≥ 24.

Exclusion Criteria:

-

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2018-07-31 (Actual); Study Completion 2018-07-31 (Actual)

PRIMARY OUTCOMES:
Weight Bearing Absolute difference between lower limbs (ΔWBA) | between the 4th and the 10th day post surgery
  Weight Bearing Absolute difference between lower limbs in kg as reported by the stabilometric platform
Weight Bearing Percentage difference between lower limbs (ΔWBP) | between the 4th and the 10th day post surgery
  Weight Bearing Percentage difference between lower limbs in % as reported by the stabilometric platform
Weight Bearing Percentage Healthy limb (WBPH) | between the 4th and the 10th day post surgery
  Weight Bearing Percentage Healthy limb in % as reported by the stabilometric platform
Weight Bearing Percentage Surgical limb (WBPS) | between the 4th and the 10th day post surgery
  Weight Bearing Percentage Surgical limb in % as reported by the stabilometric platform
Weight Bearing Absolute Healthy limb (WBAH) | between the 4th and the 10th day post surgery
  Weight Bearing Absolute Healthy limb in kg as reported by the stabilometric platform
Weight Bearing Absolute Surgical limb (WBAS) | between the 4th and the 10th day post surgery
  Weight Bearing Absolute Surgical limb in kg as reported by the stabilometric platform

SECONDARY OUTCOMES:
Mid Step Length Healthy limb (MSLH) | between the 4th and the 10th day post surgery
  Mid Step Length Healthy limb in mm as reported by the stabilometric platform
Mid Step Length Surgical limb (MSLS) | between the 4th and the 10th day post surgery
  Mid Step Length Surgical limb in mm as reported by the stabilometric platform
Sway Healthy limb (SWH) | between the 4th and the 10th day post surgery
  Sway Healthy limb in mm as reported by the stabilometric platform
Sway Surgical limb (SWS) | between the 4th and the 10th day post surgery
  Sway Surgical limb in mm as reported by the stabilometric platform
Double Support Time (DST) | between the 4th and the 10th day post surgery
  Double Support Time in ms as reported by the stabilometric platform
Numeric Rating Scale (NRS) | between the 4th and the 10th day post surgery
  Numeric Rating Scale
Six Minutes Walking Test (6MWT) | between the 4th and the 10th day post surgery
  Six Minutes Walking Test in m
World Health Organization Quality of Life Questionnaire (WHOQOL) | between the 4th and the 10th day post surgery
  World Health Organization Quality of Life Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Luca Marin, PhD, Principal Investigator — University of Pavia, Pavia, Italy
Locations (1):
- "Città di Pavia" University Hospital, Pavia, Italy, Pavia, Italy

IPD SHARING:
Plan to Share IPD: No